CLINICAL TRIAL: NCT01633034
Title: Tissue Collection for Understanding Intervertebral Disc Degeneration and Back Pain
Status: Active, not recruiting | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 10-329A
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Intervertebral Disc Degeneration; Back Pain
Keywords: intervertebral disc degeneration; back pain; spine surgery
MeSH Terms: conditions — Intervertebral Disc Degeneration; Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Intervertebral disc tissue Spinal Ligament Tissue Blood serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the research is to collect and examine spinal disc and ligament tissues to see if there are any biological markers that can be correlated with MRI images to help us learn more about causes of back pain. Spinal discs are the pillow-like cushions between the bones of the spine. They act as shock-absorbers for the spine. Spinal ligaments support the disc structure during movement.

DETAILED DESCRIPTION:
Degenerative disc disease is the most prevalent indication for spine surgery and the major source of back pain in afflicted patients. Age related degeneration of the intervertebral discs is not the exception, but the rule. Degenerative changes are associated with weakening of the disc and hypertrophy of the ligamentum flavum in the spine. The aim of this study is to determine if there are any local or systemic biomarkers that correlate with the severity of degeneration as indicated by radiological examination. To date, Imaging (XRay, MRI, CT scans) are the most widely used diagnostic tools for identifying degenerated discs. Physical changes in the disc are also associated with increased secretion and expression of inflammatory mediators in the tissue. The investigators are interested in measuring both gene and protein level changes of inflammatory mediators in degenerated discs in order to correlate these levels with imaging based indicators of degeneration. Protein level changes in the disc and ligamentum flavum have yet to be correlated with MRI-derived disc modic changes classification system. The investigators hypothesize that as the image characteristics of advancing degenerative disease increase, a corresponding change will be present in the secretion (or expression) of specific markers related to inflammatory processes in the disc. Cytokines found to be upregulated in disc tissue or ligamentum flavum will also be measured in patient's serum levels to begin developing a systemic diagnostic method for detecting disc degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Patients requiring surgery in lumbar spine region (L1-L2 to L5-S1)
3. Potential procedures: Spinal stenosis, discectomy, laminectomy, lumbar fusion, disc herniation.

Exclusion Criteria:

1. Patients requiring revision surgery in lumbar spine
2. Patients who have had a discography procedure performed at the same disc level as the one being operated on.
3. Known inflammatory conditions- Rheumatoid arthritis, Osteomyelitis, Discitis, Gout, Ankylosing spondylitis, and other infections.
4. Oncologic conditions- any history of cancer of any type.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who meet inclusion criteria will be recruited from the patients undergoing surgery at The North Shore University Hospital and at Lenox Hill Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Inflammatory profile | At surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Levine, MD, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - North Shore University Hospital, Manhasset, New York
  - Lenox Hill Hospital, Manhattan, New York

IPD SHARING:
Plan to Share IPD: No